CLINICAL TRIAL: NCT01402713
Title: Randomized, Double Blind, Multicenter, Phase II/III Study to Evaluate the Effectiveness(Immunogenicity) and Safety of 'GC1107' Administered Intramuscularly in Healthy Children
Brief Title: To Evaluate the Effectiveness(Immunogenicity) and Safety of 'GC1107' Administered Intramuscularly in Healthy Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GC1107_P2/3
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- GC1107-T5.0 (Experimental): Dosage: 0.5ml
  Interventions: Biological: GC1107
- GC1107-T7.5 (Experimental): Dosage: 0.5ml
  Interventions: Biological: GC1107
- TD_PUR INJ /SK Td vaccine (Active Comparator): The name: step 1(phase 2)-SK Td vaccine step 2(phase 3)-TD_PUR INJ Dosage: 0.5ml
  Interventions: Biological: TD_PUR INJ / SK Td vaccine

INTERVENTIONS:
Biological: GC1107 — GC1107-T5.0: low dose, GC1107-T7.5: high dose
  Arms: GC1107-T5.0; GC1107-T7.5
Biological: TD_PUR INJ / SK Td vaccine — step 1(phase 2)-TD_PUR INJ step 2(phase 3)-SK Td vaccine
  Arms: TD_PUR INJ /SK Td vaccine

SUMMARY:
The purpose of this study is to evaluate the effectiveness(immunogenicity) and safety of 'GC1107' administered intramuscularly in healthy children

DETAILED DESCRIPTION:
Randomized, double blind, multicenter, phase Ⅱ/Ⅲ study

ELIGIBILITY:
Inclusion Criteria:

* healthy Korean children(age: 10 ~ 17)

  * In the case of step1 (for step 1) 11~12 years
* who got the basic vaccination(5 times vaccination of diphtheria and tetanus until 6 years old.)
* Subjects willing to provide written informed consent and able to comply with the requirements for the study or informed consent was obtained from the subject's legal guardian

Exclusion Criteria:

* Subjects with antitoxin of diphtheria and tetanus ≥1.0IU/mL (ELISA)

  * only applicable in step 1
* subjects who have not recovered from the acute disease within 2 weeks
* who has experienced the temporary platelet decrease or has the medical history of neurologic complication
* who has the medical history of allergic disease related to the components of investigational drug
* who has experienced the severe adverse events for the diphtheria and tetanus vaccination
* who got the vaccination of diphtheria and tetanus within 5 years
* who has not recovered from the acute disease within 2 weeks
* who got the treatment of blood product within 3 months
* who got the immunoglobulin should have the wash-out period
* who be infected from the diphtheria and tetanus
* Subjects who are scheduled to participate in other clinical trial studies during the study.
* Current participation in a clinical study involving any other drugs including vaccine within 4 weeks of enrollment of the study vaccine.
* Subjects who have participated in any other clinical trials within 4 weeks of the administration of the study
* Subject who have received adrenocortical hormones or immunosuppressive drug within 4weeks of enrollment
* Subjects with a history of chronic disease obstacles to the study.
* Subjects who have episode of acute febrile (at least 37.5) after injection of vaccine during the study
* Subject who have plan of operation during the study.
* Individuals with other clinically significant medical or psychological condition who are considered by the investigator to be ineligible for the study.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 311 (Actual)
Dates: Start 2011-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Step I-the seroprotection rate of diphtheria and tetanus | 28 days
  Number of participants after vaccination as a measure of the effectiveness
Step II-to assess noninferior of diphtheria and tetanus | 28 Days

SECONDARY OUTCOMES:
StepI-GMT of diphtheria and tetanus | 28 days
Step I-safety assessment-solicited adverse event | 42 days
Step II-GMT of diphtheria and tetanus | 28 days
Step II-safety assessment-solicited adverse event | 28 days
Step II- Boosting response of diphtheria and tetanus | 28

CONTACTS AND LOCATIONS:
Overall Officials: JinHan Kang, MD, Principal Investigator — Seol St. Mary's Hospital
Locations (1):
- The catholic university of Korea, Seoul st. mary's hospital, Banpo-dong, Seoul, South Korea